CLINICAL TRIAL: NCT01360138
Title: Advantages of the Paramedian Approach for Cervical Epidural Steroid Injections: A Clinical Comparison in Cervical Epidural Pressure Changes Between Midline and Paramedian Approaches
Brief Title: A Clinical Comparison in Cervical Epidural Pressure Changes Between Midline and Paramedian Approaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Clinical Research Institute Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jymoon0901
Record Dates: First submitted 2011-05-09; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Herniated Nucleus Pulposus; Whiplash Injury
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midline approach (Active Comparator): cervical epidural steroid injection with 18G Touhy epidural needle by midline approach
  Interventions: Procedure: Cervical epidural steroid injection
- paramedian approach (Active Comparator): cervical epidural steroid injection with 18G Touhy epidural needle by paramedian approach
  Interventions: Procedure: Cervical epidural steroid injection

INTERVENTIONS:
Procedure: Cervical epidural steroid injection — cervical epidural steroid injection with a solution (5 ml) containing 10 mg triamcinolone acetonide suspension, 1.5 ml of 0.75% levobupivacaine hydrochloride, and 3.5 ml of normal saline (0.9% NaCl)

SUMMARY:
Ligamentum flavum in the cervical region is thin or not fused at the midline. The investigators inferred that the size and elasticity of the ligamentum flavum, in combination with mildline appraoch, the gaps could be responsible for a failure to recognize a LOR in some patients. If so, the investigators hypothesized that the paramedian approach would be advantageous for finding cervical epidural space more easily during cervical epidural steroid injections (CESIs).

DETAILED DESCRIPTION:
Ligamentum flavum in the cervical region is thin or not fused at the midline. The distinct elastic resistance offered by the ligamentum flavum before entering the epidural space when using the loss of resistance (LOR) technique may be blunted or even absent. The investigators inferred that the size and elasticity of the ligamentum flavum, in combination with mildline appraoch, the gaps could be responsible for a failure to recognize a LOR in some patients. If so, the investigators hypothesized that the paramedian approach would be advantageous for finding cervical epidural space more easily during cervical epidural steroid injections (CESIs). Therefore, the investigators randomly divide our patients into 2 groups; the midline approach group and the paramedian group. Then, the investigators examine the patterns of the pressure changes at the moment of a puncture of the ligamentum flavum during CESIs.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80 yr
* Cervical radicular pain caused by herniated nucleus pulposus, spinal steonosis, or other conditions, including herpes zoster-associated pain and whiplash injury for more than 3 months
* Pain intensity > 4 of maximum 10 NRS
* Failure to improve with conservative treatment
* Cervical epidural location of needle confirmed by the fluoroscopic images

Exclusion Criteria:

* Acute infection
* Patient refusal
* Previous cervical spine surgery
* Structural spinal deformities or A space-occupying epidural mass
* Rapidly worsening pain, numbness, weakness, hyperreflexia, changes in bladder function, and other neurological symptoms that should prompt a reevaluation and surgical evaluation
* Pregnancy
* Allergy to contrast media or drugs to be used in the procedure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
precipitous decrease | It will be measured at the moment of puncture of ligamentum flavum during interventional procedure, then participants will be followed for the duration of hospital stay, an expected average of 1 hour.
  Existence of the precipitous decrease in pressure at the moment of entering the cervical epidural space (exist or not)

SECONDARY OUTCOMES:
popping sensation | It will be measured at the moment of puncture of ligamentum flavum during interventional procedure, then participants will be followed for the duration of hospital stay, an expected average of 1 hour.
  Existence of the tactile sensation of give by pain experts (exist or not)
spreading levels of dye according to dye volume | It will be measured during interventional procedure, then participants will be followed for the duration of hospital stay, an expected average of 1 hour.
  Dye Volume / Dye Spreading Level after injection of 0.5 cc contrast dye, then check the spreading level such as the number of vertebral body and unilateral or bilateral spreading
cervical epidural pressure | It will be measured during interventional procedure, then participants will be followed for the duration of hospital stay, an expected average of 1 hour.
  The bevel of the needle is considered to have entered the epidural space when a typical waveform is observed, which consists of small cardiac oscillations superimposed on greater respiratory oscillations. The needle is then held immobile in the epidural space for 120 s to allow the epidural pressure to stabilize, and CEP is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea